CLINICAL TRIAL: NCT06227455
Title: Efficacy of Custom-made Zirconia Sheet Versus Polytetrafluoroethylene as a Non-resorbable Barrier in Maxillary Alveolar Ridge Augmentation
Brief Title: Efficacy of Customized Zirconia Sheet vs PTFE as a Non-resorbable Barrier in Maxillary Alveolar Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A02030123
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Alveolar Ridge Augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ti PTFE (Sham Comparator): TI PTFE is pre-bent and adapted over a 3D printed model for the alveolar defect area after virtual augmentation then used intra-operative over the mixture of Autogenous and xenograft particles.
  Interventions: Procedure: Maxillary alveolar ridge augmentation
- Customized zirconia Barrier (Active Comparator): After virtual augmentation of the defect area, a customized 3D zirconia barrier is designed on a specialized software (Autodesk Meshmixer). The exported STL file of the designed barrier is milled and sterilized. Intra-operatively, the initial try-in of the zirconia barrier is done to allow for adjustment and ensuring a proper fit and tension-free primary closure.
  Interventions: Procedure: Maxillary alveolar ridge augmentation

INTERVENTIONS:
Procedure: Maxillary alveolar ridge augmentation — The surgical procedure involves careful flap reflection, autogenous graft harvesting, and placement and fixation of the barriers over mixture of Autogenous graft and xenograft particles.

SUMMARY:
The goal of this clinical trial is comparing the efficacy of custom-made zirconia sheet versus Polytetrafluoroethylene as a non-resorbable barrier in maxillary alveolar ridge augmentation. The main question it aims to answer are:

1. Is custom made zirconia sheets are valuable as a non-resorbable membrane in guided bone regeneration?
2. Does it have any adverse effects on the surrounding tissue?
3. the accuracy of using two software in the designing of the zircon membrane?

   * Participants will be selected according to the inclusion criteria of the study, having a defect in the upper jaw that prevent rehabilitation of the jaw.
   * Participant will undergo a surgical procedure for placement of bone graft and the non-resorbable membrane.

Researchers will compare between two groups which differ only in the used membrane. a group where the researchers will place custom made zirconia sheet versus a group where the researchers will place Polytetrafluoroethylene.

DETAILED DESCRIPTION:
The study protocol demonstrates a comprehensive approach to alveolar ridge augmentation for implant placement. By utilizing 3D patient individualized zirconia barriers and TI PTFE (Titanium Reinforced Polytetrafluoroethylene) membranes, the researchers aim to compare the efficacy of these techniques in achieving successful bone gain. The preoperative evaluation, including medical history, physical examination, and CBCT, ensures that patients meet the inclusion criteria and allows for accurate planning and design of the barriers. The use of specialized software for barrier design and a computer-aided milling machine for fabrication further enhances the precision and customization of the barriers. Sterilization procedures are meticulously outlined, ensuring the safety and effectiveness of the zirconia barriers.

The surgical procedure involves careful flap reflection, autogenous graft harvesting, and placement and fixation of the barriers over mixture of Autogenous graft and xenograft particles . In Group I, the TI PTFE membrane is shaped and pre-bent on a 3D printed augmented model then fixed over the graft and alveolar defect to adapt to the alveolar defect, providing a protective barrier for the graft. In Group II, the initial try-in of the zirconia barrier allows for adjustments to ensure a proper fit and tension-free primary closure. Finally the zirconia membrane is placed over the harvested bone in the recipient site. Both barriers are fixed with bone screws at well marked computer guided positions ensuring the safety of neighboring teeth and vital structures.

The evaluation process involves cone beam CT and clinical assessment at specific intervals to evaluate bone gain, soft tissue inflammation, infection, and dehiscence. The use of 3D models and software allows for accurate volumetric analysis and measurement of the alveolar ridge dimensions, providing valuable data for evaluation.

In conclusion, this study protocol demonstrates a meticulous and comprehensive approach to alveolar ridge augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be free from any relevant systemic disease that would contraindicate surgical intervention or affect bone healing.
* Patients with single or multiple missing teeth with vertical alveolar defect or severe horizontal defect or both types of defects, preventing placement of any implant or prosthetic appliance in maxilla.
* Clinically apparent increase in interarch space relative to the adjacent alveolar teeth.

Exclusion Criteria:

* History of uncontrolled medical disorders.
* History of systemic diseases or medication that alter bone metabolism.
* Poor oral hygiene.
* Heavy smoker (more than ten cigarettes/day) or alcoholic patients.
* Chemotherapy or Radiation therapy to the head and neck region in the 12 months prior to the proposed therapy.
* Patients currently on or with a history of bisphosphonate therapy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Bone volume in cubic millimeters | First postoperative week
  Volume of the gained bone is assessed by cone-beam computed tomography (CBCT)
Bone volume in cubic millimeters | Sixth postoperative month
  Volume of the gained bone is assessed by cone-beam computed tomography (CBCT)

SECONDARY OUTCOMES:
Clinical examination | Sixth postoperative months
  Patients are examined for any cardinal sign of inflammation (Positive/negative)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Addakahlyia, Egypt

REFERENCES:
- [Derived] Sakr MI, Salem AS, Yaseen AA, Tawfik MA, Mansour NA. Early postoperative evaluation of an open-source digital workflow for designing custom-made zirconia membranes in maxillary guided bone regeneration. BMC Oral Health. 2025 Jul 18;25(1):1200. doi: 10.1186/s12903-025-06592-0. PMID 40682045